CLINICAL TRIAL: NCT03712930
Title: A Phase 2, Open-Label, Single-Arm Study of BGB-290 (BGB-290) for the Treatment of Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC) With Homologous Recombination Deficiency (HRD)
Brief Title: Treatment of Metastatic Castration-Resistant Prostate Cancer With Homologous Recombination Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to revisit the development approach for prostate cancer.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-290-202; 2018-002587-28 (EudraCT Number)
Record Dates: First submitted 2018-10-11; First posted 2018-10-19 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC); Homologous Recombination Deficiency (HRD)
MeSH Terms: interventions — pamiparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pamiparib (Experimental): Participants will receive pamiparib for a period up to 1 year
  Interventions: Drug: Pamiparib

INTERVENTIONS:
Drug: Pamiparib — 60 mg orally twice daily (BID)
  Other Names: BGB-290

SUMMARY:
This study is designed to evaluate the efficacy of pamiparib in participants with metastatic castration-resistant prostate cancer (mCRPC) positive for circulating tumor cells (CTC) with homologous recombination deficiency (CTC-HRD). All participants will receive pamiparib. The purpose of this study is to demonstrate that pamiparib will improve Objective Response Rate (ORR) and Prostate-Specific Antigen (PSA) response rate

DETAILED DESCRIPTION:
This is a global, Phase 2, open-label study of pamiparib in approximately 100 participants with metastatic castration-resistant prostate cancer (mCRPC) positive for circulating tumor cells (CTC) with homologous recombination deficiency (CTC-HRD). Participants in Cohort 1 will include 50 mCRPC participants with CTC-HRD-positive, measurable metastatic disease (soft tissue with/without bone lesions), and positive BRCA1/2 mutation or negative/unknown BRCA1/2 mutation. Cohort 2 will include 30 mCRPC CTC-HRD positive participants with bone metastasis only and positive or negative/unknown BRCA1/2. Cohort 3 and 4 will include 20 mCRPC CTC-HRD negative/unknown participants with BRCA1/2 positive mutations, metastatic disease (measurable soft tissue with/without bone), and bone only. Participants will undergo PSA level assessments approximately every 4 weeks as well as tumor assessments every 8 weeks for 24 weeks and the every 12 weeks, or as clinically indicated. Administration of pamiparib will continue until disease progression, unacceptable toxicity, death or another discontinuation criterion is met.

ELIGIBILITY:
Key Inclusion Criteria:

* Men (≥ 18 years of age) with histologically or cytologically confirmed adenocarcinoma or poorly differentiated adenocarcinoma of the prostate without neuroendocrine differentiation with HRD deficiency by CTC-HRD assay and/or deleterious germline or somatic mutation in BRCA1 or BRCA2; mCRPC measurable disease and/or bone disease. • PSA progression with ≥ 3 rising PSA levels with ≥ 1 week between determinations and a screening PSA ≥ 2 μg/L (2 ng/mL).
* Must be surgically or medically castrated with serum testosterone levels of ≤1.73 nmol/L (50 ng/dL), must have received ≥ 1 prior androgen receptor-targeted therapy, and must have received ≥ 1 taxane-based therapy.
* mCRPC with 1 or 2 of the following:
* Measurable disease per RECIST v1.1
* Bone disease
* CTC-HRD+ or BRCA1/2 mutation
* PSA progression (PCWG3 criteria)
* ≥1 androgen receptor-targeted therapy (eg, abiraterone acetate/prednisone or enzalutamide) for mCRPC with progressive disease
* ≥1 taxane for metastatic prostate cancer

Key Exclusion Criteria:

* Chemotherapy, hormonal therapy, biologic therapy, radionuclide therapy, immunotherapy, investigational agent, anticancer Chinese medicine, or herbal remedies ≤ 5 half-lives if the half-life is known, ≤ 14 days if not known, before start of study treatment
* Continued treatment with a bisphosphonate or denosumab is allowed, if administered at a stable dose > 28 days before start of study treatment
* Radiotherapy ≤ 21 days (≤ 14 days, if single fraction of radiotherapy) before start of study treatment

Prior treatment for prostate cancer with any of the following:

* poly ADP ribose polymerase (PARP) inhibitor
* Platinum
* Cyclophosphamide
* Mitoxantrone

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (9):
- United States (3):
  - University Cancer and Blood Center, Athens, Georgia
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - University of Washington, Seattle, Washington
- Australia (4):
  - Gosford Hospital, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Icon Cancer Care Foundation, South Brisbane, Queensland
- Pan American Oncology Trials, LLC, Rio Piedras, Puerto Rico
- L Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen subjects were screened; 5 subjects failed screening and 13 subjects were dosed.
Pre-assignment Details: All subjects enrolled had unknown BRCA1/2 status at study entry and were assigned to cohorts 1B or 2B; there were no subjects known to be BRCA1/2 positive at enrollment.
Groups:
- Pamiparib: Participants received 60 mg pamiparib orally twice daily
Period: Overall Study
Arm/Group | Pamiparib
Started | 13
Completed | 0
Not Completed | 13
Not completed — Death | 7
Not completed — Physician Decision | 1
Not completed — Study Terminated by Sponsor | 3
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native, White | 1
  Race: White | 7
  Race: Not Reported | 1
  Race: Unknown | 3
  Race: Other | 1
  Ethnicity: Not Hispanic or Latino | 7
  Hispanic or Latino | 3
  Not Reported/Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Determined by Independent Review Committee
Description: ORR is the percentage of participants with a best objective response of complete response (CR) or partial response (PR) confirmed at a subsequent timepoint ≥ 4 weeks later by an Independent Review Committee (IRC).
Time Frame: Up to 1 year and 6 months
Population: Efficacy-Evaluable Analysis Set: includes all participants in the Safety Analysis Set who had measurable disease at baseline and at least 1 post-baseline tumor assessment, unless they permanently discontinue pamiparib or the study early due to clinical progression or death before tumor assessment. Participants with available data were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 12
Percentage of participants | 0

2. Primary Outcome: Prostate-Specific Antigen (PSA) Response Rate
Description: PSA response rate is defined as the percentage of participants with PSA decline ≥ 50% from baseline [confirmed by a second PSA value ≥ 3 weeks later] for CTC-HRD-positive participants with or without measurable disease.
Time Frame: Up to 1 year and 6 months
Population: PSA-Evaluable Analysis Set: includes all participants in the Safety Analysis Set with ≥3 rising PSA levels with ≥ 1 week between determinations and screening PSA ≥ 2 μg/L) and who had at least 1 post-baseline PSA measurement unless they permanently discontinue pamiparib or the study early due to clinical progression or death before completed PSA assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Percentage of participants | 0

3. Secondary Outcome: Duration of Response (DOR) by IRC
Description: DOR is defined as the time from the date of the earliest documented CR or PR (that is subsequently confirmed) to radiographic disease progression or death due to any cause, whichever occurs first.
Time Frame: Up to 1 year and 7 months
Population: as for outcome 1
Measure: Number; unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 12
Months | NA — No confirmed CR/PR. Duration of Response is not applicable.

4. Secondary Outcome: Objective Response Rate by Investigator
Description: ORR is the percentage of participants with a best objective response of complete response (CR) or partial response (PR) confirmed at a subsequent timepoint ≥ 4 weeks later by the investigator.
Time Frame: Up to 1 year and 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 12
Percentage of participants | 0

5. Secondary Outcome: Time to Objective Response by Investigator
Description: Time to objective response is defined as the time from the date of the first dose of study drug to the first documented confirmed response of CR or PR assessed by the investigator and summarized for participants who have achieved a confirmed objective response.
Time Frame: Up to 1 year and 6 months
Population: as for outcome 1
Measure: Number; unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 12
Months | NA — No participants with confirmed CR/PR. Time to response is not applicable.

6. Secondary Outcome: Clinical Benefit Rate By Investigator
Description: Clinical Benefit Rate is the percentage of participants who achieved confirmed CR, PR, or SD or NON-CR/NON-PD. The minimum interval for confirmed CR and PR is 4 weeks and the measurement of SD or NON-CR/NON-PD is 7 weeks after first dose date.
Time Frame: Up to 1 year and 6 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 12
Percentage of participants | 25

7. Secondary Outcome: Time to PSA Response
Description: Time to PSA response is defined as the time from the date of the first dose of study drug to the first PSA decline ≥ 50% that is subsequently confirmed. Assessments are summarized for participants who have achieved a confirmed PSA response.
Time Frame: Up to 1 year and 6 months
Population: PSA-Evaluable Analysis Set: includes all participants in the Safety Analysis Set with ≥3 rising PSA levels with ≥ 1 week between determinations and screening PSA ≥ 2 μg/L and who had at least 1 post-baseline PSA measurement, unless they permanently discontinue pamiparib or the study early due to clinical progression or death before completed PSA assessment.
Measure: Number; unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Months | NA — Number of participants with PSA response is 0. Time to PSA response is not applicable.

8. Secondary Outcome: Duration of PSA Response
Description: Duration of PSA response is defined as the time from the date of the earliest documented PSA response (that is subsequently confirmed) to PSA progression or death due to any cause, whichever occurs first. PSA progression is defined as a ≥ 25% increase in PSA with an absolute increase of ≥ 2 μg/L above the nadir (or above the baseline for participants with no PSA decline) after12 weeks, confirmed by a second value ≥ 3 weeks later. The nadir is defined as the lowest value at or after baseline.
Time Frame: Up to 1 year and 7 months
Population: PSA-Evaluable Analysis Set: includes all participants in the Safety Analysis Set with ≥3 rising PSA levels with ≥ 1 week between determinations and screening PSA ≥ 2 μg/L) and who had at least 1 post-baseline PSA measurement, unless they permanently discontinue pamiparib or the study early due to clinical progression or death before completed PSA assessment.
Measure: Number; unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Months | NA — The number of participants with PSA Response is 0. Duration of PSA response is not applicable.

9. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression is defined as the time from the date of the first dose of study drug to a ≥ 25% increase in PSA with an absolute increase of ≥ 2 ng/mL above the nadir (or above the baseline for participants with no PSA decline) after 12 weeks, confirmed by a second value ≥ 3 weeks later. Death for the participants with no PSA progression is also considered as an event.
Time Frame: Up to 1 year and 7 months
Population: Safety Analysis Set : includes all participants enrolled into the study who received any dose of pamiparib.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Months | 3.13 (1.533)

10. Secondary Outcome: Time to Symptomatic Skeletal Event
Description: Time to symptomatic skeletal event (SSE) is defined as time from the date of the first dose of study drug to the first symptomatic fracture, radiation or surgery to bone, or spinal cord compression.
Time Frame: Up to 1 year and 7 months
Population: Safety Analysis Set: includes all participants enrolled in the study who received any dose of pamiparib
Measure: Number; unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Months | NA — No participants had SSE

11. Secondary Outcome: Radiographic Progression-Free Survival by IRC
Description: Radiographic progression-free survival is defined as the time from the date of the first dose of study drug to radiographic disease progression by IRC or death due to any cause, whichever occurs first.
Time Frame: Up to 1 year and 7 months
Population: Safety Analysis Set : includes all participants enrolled in the study who received any dose of pamiparib
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Months | 2.6 [1.5 to 3.7]

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of the first dose of study drug to death due to any cause.
Time Frame: Up to 1 year and 7 months
Population: Safety Analysis Set: includes all participants enrolled in the study who received any dose of pamiparib
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
Months | 5.8 [1.6 to 5.9]

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events Graded According to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03
Time Frame: From the date of first Pamiparib dose until 30 days after the last dose or initiation of new anti-cancer therapy, whichever occurs first. (Up to 1 year and 7 months)
Population: Safety Analysis Set: includes all participants enrolled in the study who received any dose of pamiparib
Measure: Number; unit: number of participants
Arm/Group | Pamiparib
Number analyzed (Participants) | 13
number of participants
  Participants with at Least One TEAE | 13
  Grade 3 or Higher | 11
  Serious | 6
  Leading to Death | 1
  Leading to Treatment Discontinuation | 3
  Leading to Dose Modification | 11
  Leading to Dose Interruption | 9
  Leading to Dose Reduction | 5
  Treatment Related TEAEs | 11
  Treatment Related Grade 3 or Higher | 7
  Treatment Related Serious | 1
  Treatment Related Leading to Death | 0
  Treatment Related Leading to Treatment Discontinuation | 3
  Treatment Related Leading to Dose Modification | 7
  Treatment Related Leading to Dose Interruption | 6
  Treatment Related Leading to Dose Reduction | 3

ADVERSE EVENTS:
Time Frame: From the date of first dose of Pamiparib until 30 days after the last dose or initiation of new anti-cancer therapy, whichever occurs first (up to approximately 1 year and 7 months)
Arm/Group | Pamiparib
All-Cause Mortality (participants affected / at risk) | 9/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pamiparib (N=13)
Pyrexia (General disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Peripheral swelling (General disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pamiparib (N=13)
Anaemia (Blood and lymphatic system disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 6
Fatigue (General disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Weight decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Asthenia (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Constipation (Gastrointestinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Headache (Nervous system disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Orbital oedema (Eye disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Platelet count decreased (Investigations) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectal tenesmus (Gastrointestinal disorders) | 1
Taste disorder (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03712930/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT03712930/SAP_001.pdf